CLINICAL TRIAL: NCT01651481
Title: Open-label, Randomized, Single Dose Crossover Study to Evaluate the Pharmacokinetics and Safety of Singulair (10 mg) and Xyzal (5 mg) in Free Combination and Fixed-dose Combination as HCP1102 in Healthy Male Volunteers
Brief Title: Study to Evaluate the Pharmacokinetics and Safety of Singulair and Xyzal in Free Combination and Fixed-dose Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-MOLZ-102
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Rhinitis
Keywords: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — montelukast; levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TR (Experimental): HCP1102(Singulair and Xyzal combination tablet) -> coadministration of Singulair and Xyzal
  Interventions: Drug: HCP1102; Drug: Singulair and Xyzal
- RT (Experimental): coadministration of Singulair and Xyzal -> HCP1102(Singulair and Xyzal combination tablet)
  Interventions: Drug: HCP1102; Drug: Singulair and Xyzal

INTERVENTIONS:
Drug: HCP1102
  Other Names: Singulair and Xyzal combination tablet
Drug: Singulair and Xyzal
  Other Names: coadministration of Singulair and Xyzal

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of Singulair (10 mg) and Xyzal (5 mg) in free combination and fixed-dose combination as HCP1102

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Age between 20 and 55
* Signed informed consent

Exclusion Criteria:

* Has a history of hypersensitivity to IP ingredients
* Hypotension or hypertension
* Has a history of acute infection within 14 days of screening

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
AUClast | 0-34hr
Cmax | 0-34hr

SECONDARY OUTCOMES:
tmax | 0-34hr
AUCinf | 0-34hr
t1/2 | 0-34hr

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea